CLINICAL TRIAL: NCT04298528
Title: A Prospective, Randomized, Double Blind Trial Comparing Dronabinol to a Placebo in the Management of Post-operative Pain in Total Joint Arthroplasty
Brief Title: A RCT Comparing Dronabinol to a Placebo for Post-operative Pain in Total Joint Arthroplasty
Acronym: dronabinol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Principal Investigator, Jason Jennings, Orthopedic Surgeon, Colorado Joint Replacement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1554107
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dronabinol; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dronabinol (Experimental): Patient will be directed to take 2.5mg of Study Drug 2 times a day for 4 weeks. Patient is blinded as to whether or not this is Dronabinol.
  Interventions: Drug: Dronabinol
- placebo (Placebo Comparator): Patient will be directed to take 2.5mg of Study Drug 2 times a day for 4 weeks. Patient is blinded as to whether or not this is Dronabinol.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dronabinol — 2.5mg 2 times a day for 30 days after total knee replacement
  Other Names: Marinol
  Arms: dronabinol
Other: Placebo — 2 times a day for 30 days after total knee replacement
  Other Names: Lactose
  Arms: placebo

SUMMARY:
The primary purpose of this study was to determine if cannabinoid use decreases narcotic consumption in patients undergoing total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Subjects enrolled will be randomized into one of two groups either receiving the study drug or a placebo and will be followed for the first 6 weeks with regards to outcomes data.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent from
* Stated willingness to comply with all study procedures and availability to attend all required visits for the duration of the study.
* Male or Female
* Age 21-75
* Unilateral total knee arthroplasty at Colorado Joint Replacement
* All individuals will be screened for drug use (including cannabis) at their preoperative appointment
* Ability to take oral medication and be willing to adhere to the dronabinol regimen
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

* Narcotic use in the past 6 weeks
* Regular cannabis use in the past 3 months
* Major depression or anxiety disorders
* Documented psychiatric illness (e.g. bipolar, schizophrenia)
* Seizure disorder
* Current or previous history of drug and alcohol abuse
* Known allergic reactions to components of dronabinol
* Tobacco use in the past 90 days
* Treatment with another investigational drug
* Patients that cannot receive spinal anesthesia
* Patients that cannot receive the standardized multimodal pain medications (i.e. Tylenol, gabapentin and meloxicam)
* Patients that are not able to go home after leaving the hospital and require a short term rehabilitation facility

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
Morphine Equivalence | 30 day's post operative
  Morphine Equivalence of pain medication used after a total knee replacement

SECONDARY OUTCOMES:
Nausea | 30 day's post operative
  Patients post operative nausea will be collected as none/mild/moderate/severe
Defense and Veterans Pain Scale | 30 day's post operative
  Patients will keep a pain log after their joint replacement on a scale of 0 - 10
The Pittsburgh Sleep Quality Index | 4 weeks and 6 weeks post operative
  To monitor sleeping habits
Knee Society Score | 4 weeks post operative
  Patient reported outcome
KOOS-12 Knee Survey | 6 weeks post operative
  Patient reported outcome
The Veterans Rand 12-Item Health Survey | 6 weeks post operative
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Jennings, MD DPT, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hannon CP, Calkins TE, Li J, Culvern C, Darrith B, Nam D, Gerlinger TL, Buvanendran A, Della Valle CJ. The James A. Rand Young Investigator's Award: Large Opioid Prescriptions Are Unnecessary After Total Joint Arthroplasty: A Randomized Controlled Trial. J Arthroplasty. 2019 Jul;34(7S):S4-S10. doi: 10.1016/j.arth.2019.01.065. Epub 2019 Feb 4. PMID 30799266
- [Background] Jennings JM, Williams MA, Levy DL, Johnson RM, Eschen CL, Dennis DA. Has Self-reported Marijuana Use Changed in Patients Undergoing Total Joint Arthroplasty After the Legalization of Marijuana? Clin Orthop Relat Res. 2019 Jan;477(1):95-100. doi: 10.1097/CORR.0000000000000339. PMID 30794232
- [Background] Hickernell TR, Lakra A, Berg A, Cooper HJ, Geller JA, Shah RP. Should Cannabinoids Be Added to Multimodal Pain Regimens After Total Hip and Knee Arthroplasty? J Arthroplasty. 2018 Dec;33(12):3637-3641. doi: 10.1016/j.arth.2018.07.027. Epub 2018 Aug 3. PMID 30170713
- [Background] Hayes MJ, Brown MS. Legalization of medical marijuana and incidence of opioid mortality. JAMA Intern Med. 2014 Oct;174(10):1673-4. doi: 10.1001/jamainternmed.2014.2716. No abstract available. PMID 25156148
- [Background] Heng M, McTague MF, Lucas RC, Harris MB, Vrahas MS, Weaver MJ. Patient Perceptions of the Use of Medical Marijuana in the Treatment of Pain After Musculoskeletal Trauma: A Survey of Patients at 2 Trauma Centers in Massachusetts. J Orthop Trauma. 2018 Jan;32(1):e25-e30. doi: 10.1097/BOT.0000000000001002. PMID 29257781
- [Background] Khelemsky Y, Goldberg AT, Hurd YL, Winkel G, Ninh A, Qian L, Oprescu A, Ciccone J, Katz DJ. Perioperative Patient Beliefs Regarding Potential Effectiveness of Marijuana (Cannabinoids) for Treatment of Pain: A Prospective Population Survey. Reg Anesth Pain Med. 2017 Sep/Oct;42(5):652-659. doi: 10.1097/AAP.0000000000000654. PMID 28796754
- [Background] Chan MH, Knoepke CE, Cole ML, McKinnon J, Matlock DD. Colorado Medical Students' Attitudes and Beliefs About Marijuana. J Gen Intern Med. 2017 Apr;32(4):458-463. doi: 10.1007/s11606-016-3957-y. Epub 2017 Jan 17. PMID 28097606
- [Background] Cancienne JM, Patel KJ, Browne JA, Werner BC. Narcotic Use and Total Knee Arthroplasty. J Arthroplasty. 2018 Jan;33(1):113-118. doi: 10.1016/j.arth.2017.08.006. Epub 2017 Aug 17. PMID 28887020
- [Background] Menendez ME, Ring D, Bateman BT. Preoperative Opioid Misuse is Associated With Increased Morbidity and Mortality After Elective Orthopaedic Surgery. Clin Orthop Relat Res. 2015 Jul;473(7):2402-12. doi: 10.1007/s11999-015-4173-5. Epub 2015 Feb 19. PMID 25694266
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Di Marzo V, Bifulco M, De Petrocellis L. The endocannabinoid system and its therapeutic exploitation. Nat Rev Drug Discov. 2004 Sep;3(9):771-84. doi: 10.1038/nrd1495. PMID 15340387
- [Background] Fitzcharles MA, Hauser W. Cannabinoids in the Management of Musculoskeletal or Rheumatic Diseases. Curr Rheumatol Rep. 2016 Dec;18(12):76. doi: 10.1007/s11926-016-0625-5. PMID 27832442